CLINICAL TRIAL: NCT00118469
Title: Parent Psychoeducation Intervention in CBT for Depressed Latino Youth
Brief Title: Parent Psychoeducation and Cognitive Behavior Therapy for Latino Adolescents With Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: R01MH067893 (NIH); DSIR 84-CTS
Record Dates: First submitted 2005-07-06; First posted 2005-07-11 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-02

CONDITIONS: Depression
Keywords: Adolescent; CBT; Parents
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Psychoeducation
Behavioral: Cognitive behavior therapy

SUMMARY:
This study will determine the effectiveness of adding a parent-involved intervention to cognitive behavior therapy in reducing depressive symptoms among Latino adolescents with depression.

DETAILED DESCRIPTION:
Adolescent depression can have a devastating impact on social, emotional, and family functioning. Cognitive behavior therapy (CBT) is the most common treatment for depression; however, not all patients respond adequately to CBT. In addition, data on the effects of CBT among ethnic minorities are limited. Because Latinos are the largest minority group in the United States, the development of treatments specifically designed for depressed Latino youth are needed. This study will determine whether adding a psychoeducation intervention with parent involvement will be more effective in reducing depressive symptoms among Latino adolescents than treatment with CBT alone.

The treatment phase of this study will last 12 weeks. Participants will be randomly assigned to receive 12 weeks of either CBT alone or CBT with psychoeducation. The psychoeducation will consist of 8 sessions over the 12-week treatment period. During the sessions, participants and their parents will be given detailed information about depression and ways the condition can be treated. They will also be taught coping skills and ways to recognize a relapse. CBT sessions will take place weekly during the study. During the sessions, a therapist will work with participants to modify the behavior and thinking patterns that cause and are associated with their depressive symptoms. Both participants and their parents will undergo interviews at study start, study completion, and 3, 9, and 15 months after study completion. During the interviews, participants' depressive symptoms, school attendance, and overall functional status will be assessed. Parents' stress levels and work attendance will also be assessed. At Months 6 and 12 after study completion, participants and their parents will complete questionnaires to assess any relapses in depressive symptoms.

Study hypothesis: Active treatment with psychoeducation will be superior to no psychoeducation in reducing depression post-treatment. Because the psychoeducation intervention is designed to involve parents and thus impact other aspects of the family system, the treatment is expected to produce better outcomes in several functional domains.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depression
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Psychiatric conditions other than depression

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2004-07; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
General functioning status
family functioning
school attendance
attrition rates

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Bernal, PhD, Principal Investigator — University Center for Psychological Services and Research, University of Puerto Rico
Locations (1):
- University Center for Psychological Services and Research, University of Puerto Rico, San Juan, Puerto Rico